CLINICAL TRIAL: NCT00632411
Title: Efficacy of a Smoking Quit Line in the Military
Brief Title: Evaluating a Telephone-Based Smoking Cessation Program Among People in the Military (The AFIII Study)
Acronym: AFIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 524; R18HL053478-07A2 (NIH)
Record Dates: First submitted 2008-03-06; First posted 2008-03-10 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2016-09

CONDITIONS: Smoking; Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proactive group (Experimental): Research study staff will contact participant to initiate the program. Half of participants will be randomized to the proactive condition and the other half to the reactive conditions.
  Interventions: Drug: Nicotine Patch; Behavioral: Tobacco Quit Line Program
- Reactive group (Experimental): Participant will contact the research study staff to initiate the program.
  Interventions: Drug: Nicotine Patch; Behavioral: Tobacco Quit Line Program

INTERVENTIONS:
Drug: Nicotine Patch — Participants who smoke more than 20 cigarettes per day will use a 21-mg patch for 4 weeks, a 14-mg patch for the next 2 weeks, a 7-mg patch for the next 2 weeks, and then no patch.
  Participants who smoke between 10 to 19 cigarettes per day will use a 14-mg patch for 4 weeks, a 7-mg patch for the next 4 weeks, and then no patch.
  Participants who smoke between 5 to 9 cigarettes per day will use a 7-mg patch for 8 weeks and then no patch.
  The proactive group will be given 8 weeks of patch treatment and the reactive group will be given 2 weeks of patch treatment.
Behavioral: Tobacco Quit Line Program — Phone session 1 will focus on smoking reduction.
  Phone session 2 will focus on preparing to quit and surviving the first days as a non-smoker. A quit date will be set in 7 to 10 days. Nicotine patches will be sent to participant with detailed instructions for patch use.
  Phone session 3 will focus on the first days after the quit date.
  Phone session 4 will focus on a review of progress and challenges of quitting. Plans to manage high-risk situations will be discussed.
  Phone session 5 will focus on short-term relapse prevention.
  Phone session 6 will focus on long-term relapse prevention.

SUMMARY:
Rates of cigarette smoking in the military are high. Tobacco telephone quit lines are telephone-based services that provide information and guidance to people who want to quit smoking. This study will evaluate the effectiveness of a tobacco quit line program, in addition to nicotine replacement patches, at helping people in the military quit smoking cigarettes.

DETAILED DESCRIPTION:
Active duty military personnel are at high risk of cigarette smoking. Despite strong efforts by the Department of Defense to reduce tobacco use, rates of smoking among people in the military remain high. The military lifestyle presents unique challenges to implementing smoking cessation programs, including the high mobility of troops, remote locations, and limited access to healthcare services. Because of these challenges, many smoking cessation programs that are effective in the non-military population are often ineffective in the military population. Tobacco telephone quit lines are telephone-based tobacco cessation services that provide easy access to educational materials, referrals to local programs, and individualized telephone counseling. Because tobacco quit lines are remotely based and can fit into varying schedules at convenient times, they may be effective among people in the military. Nicotine replacement patches are another effective smoking cessation tool and can be used in addition to telephone quit lines. The purpose of this study is to evaluate the effectiveness of tobacco quit lines, in addition to nicotine replacement patches, at improving smoking cessation rates among members of the Air Force.

This study will enroll military healthcare beneficiaries who have smoked at least five cigarettes a day in the year before study entry. Participants will be randomly assigned to either a proactive group, in which study researchers will initiate contact with the participants, or a reactive group, in which participants will initiate contact with the researchers. In this six-session program, phone calls will occur at 1- to 2-week intervals over an 8-week period. The phone sessions will focus on cutting down on cigarette smoking, setting a quit date, and relapse prevention. All participants will receive nicotine replacement patches after the second session is completed. The reactive group will receive two weeks of nicotine replacement patches and the proactive group will receive 8 weeks of nicotine replacement patches. At the end of session four and 1 year later, study staff will call participants to collect information on tobacco abstinence, nicotine replacement patch use adherence, and other smoking cessation medication use.

ELIGIBILITY:
Inclusion Criteria:

* Department of Defense healthcare beneficiary
* Has smoked five or more cigarettes per day for at least 1 year before study entry
* Must be at least eighteen years old

Exclusion Criteria:

* Known allergy or sensitivity to nicotine replacement therapy
* No telephone
* Inability to understand consent procedures
* Basic Military Trainee

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1298 (Actual)
Dates: Start 2008-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Klesges, PhD, Principal Investigator — University of Tennessee Health Science Center and St. Jude Childrens' Research Hospital; Harry Lando, PhD, Principal Investigator — University of Minnesota; Gerald W. Talcott, Ph.D. Colonel (Ret.), Principal Investigator — Wilford Hall Medical Center; University of Tennessee Health Science Center
Locations (2):
- United States (2):
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Annual smoking-attributable mortality, years of potential life lost, and economic costs--United States, 1995-1999. MMWR Morb Mortal Wkly Rep. 2002 Apr 12;51(14):300-3. PMID 12002168
- [Background] Mokdad AH, Marks JS, Stroup DF, Gerberding JL. Actual causes of death in the United States, 2000. JAMA. 2004 Mar 10;291(10):1238-45. doi: 10.1001/jama.291.10.1238. PMID 15010446
- [Background] Bray RM, Hourani LL, Rae KL, al. e: Department of Defense Survey of Health Related Behaviors Among Military Personnel, in Report No. RTI/7841/006-FR, Research Triangle Park, NC, RTI International, 2003
- [Background] U.S. Department of Health and Human Services: The health consequences of smoking; a report of the surgeon general., in, Atlanta, GA, USDHHS, Centers for Disease Control and Prevention, National Center for Chronic Disease and Prevention and Health Promotion, Office on Smoking and Health, 2004
- [Background] Centers for Disease Control and Prevention (CDC). Cigarette smoking among adults--United States, 2002. MMWR Morb Mortal Wkly Rep. 2004 May 28;53(20):427-31. PMID 15163928
- [Background] Department of Defense: Tobacco use prevention strategic plan., in, Washington, D.C., Department of Defense, 1999
- [Background] Department of Defense: Smoking in DoD occupied buildings and facilities., in, Washington, DC, Department of Defense, 1977, p Instruction No. 6015.6018
- [Background] Department of Defense: Health promotion., in, Washington, D.C., Department of Defense, 1994b, pp Directive No. 1010.1010 (1010.1010 supersedes and cancels March 1011, 1986, version of Directive No. 1010.1010)
- [Background] Department of Defense: DoD food and nutrition research, development, testing, evaluation, and engineering program., in, Washington, D.C., Department of Defense, 1983, p Instruction No. 3235.3232
- [Background] Conway TL, Woodruff SI, Edwards CC, Elder JP, Hurtado SL, Hervig LK. Operation Stay Quit: evaluation of two smoking relapse prevention strategies for women after involuntary cessation during US Navy recruit training. Mil Med. 2004 Mar;169(3):236-42. doi: 10.7205/milmed.169.3.236. PMID 15080246
- [Background] Cronan TA, Conway TL, Hervig LK. Evaluation of smoking interventions in recruit training. Mil Med. 1989 Jul;154(7):371-5. PMID 2503780
- [Derived] Klesges RC, Ebbert JO, Talcott GW, Thomas F, Richey PA, Womack C, Hryshko-Mullen A, Oh J. Efficacy of a Tobacco Quitline in Active Duty Military and TRICARE Beneficiaries: A Randomized Trial. Mil Med. 2015 Aug;180(8):917-25. doi: 10.7205/MILMED-D-14-00513. PMID 26226536

RESULTS

PARTICIPANT FLOW:
Groups:
- Proactive Group: Study staff will initiate contact to conduct 6 individual counseling sessions.
  Participants will receive 8 weeks of Nicotine Replacement Therapy in the form of a patch.
- Reactive Group: Participant will initiate contact with participant to conduct 6 individual counseling sessions.
  Participants will receive 2 weeks of Nicotine Replacement Therapy in the form of a patch.
Period: Overall Study
Arm/Group | Proactive Group | Reactive Group
Started | 649 | 649
Completed | 489 | 473
Not Completed | 160 | 176

BASELINE CHARACTERISTICS:
Groups:
- Proactive Group: Research study staff will contact participant to initiate sessions.
  8 weeks of Nicotine Replacement Therapy in the form of patch will be distributed this group.
  Six sessions will be proactively delivered to the participant.
  Phone session 1 will focus on smoking reduction.
  Phone session 2 will focus on preparing to quit and surviving the first days as a non-smoker. A quit date will be set in 7 to 10 days.
  Phone session 3 will focus on the first days after the quit date.
  Phone session 4 will focus on a review of progress and challenges of quitting. Plans to manage high-risk situations will be discussed.
  Phone session 5 will focus on short-term relapse prevention.
  Phone session 6 will focus on long-term relapse prevention.
- Reactive Group: Participant will contact the research study staff to initiate sessions.
  2 weeks of Nicotine Replacement Therapy in the form of patch will be distributed this group.
  Six sessions will be delivered to the participant as long as the participant calls to initiate the sessions.
  Phone session 1 will focus on smoking reduction.
  Phone session 2 will focus on preparing to quit and surviving the first days as a non-smoker. A quit date will be set in 7 to 10 days.
  Phone session 3 will focus on the first days after the quit date.
  Phone session 4 will focus on a review of progress and challenges of quitting. Plans to manage high-risk situations will be discussed.
  Phone session 5 will focus on short-term relapse prevention.
  Phone session 6 will focus on long-term relapse prevention.
- Total: Total of all reporting groups
Arm/Group | Proactive Group | Reactive Group | Total
Number analyzed (Participants) | 649 | 649 | 1298
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 649 | 649 | 1298
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.59 (13.65) | 39.42 (13.82) | 39.50 (13.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 291 | 271 | 562
  Male | 358 | 378 | 736
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 61 | 124
  Not Hispanic or Latino | 585 | 588 | 1173
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 8 | 14
  Asian | 7 | 10 | 17
  Native Hawaiian or Other Pacific Islander | 13 | 5 | 18
  Black or African American | 85 | 75 | 160
  White | 493 | 509 | 1002
  More than one race | 24 | 24 | 48
  Unknown or Not Reported | 21 | 18 | 39
Region of Enrollment [Number; unit: participants]
  United States | 649 | 649 | 1298

OUTCOME MEASURES:

1. Primary Outcome: Continuous Abstinence
Description: No cigarette smoking since two weeks after the target quit date.
Time Frame: Measured at Year 1
Population: Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Proactive Group | Reactive Group
Number analyzed (Participants) | 521 | 529
Participants | 173 | 136

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Proactive Group | Reactive Group
Serious Adverse Events (participants affected / at risk) | 16/649 | 6/649
Other Adverse Events (participants affected / at risk) | 307/649 | 98/649
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proactive Group (N=649) | Reactive Group (N=649)
Hospitalization (Surgical and medical procedures) | 16 (16) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proactive Group (N=649) | Reactive Group (N=649)
Headache (General disorders) | 14 (14) | 4 (4)
Skin Rash (Injury, poisoning and procedural complications) | 88 (88) | 26 (26)
Sleep Disturbance (Injury, poisoning and procedural complications) | 64 (64) | 19 (19)
Respiratory illness/ Sinus/ Sore throat/ Cold/Flu/Seasonal allergies (Respiratory, thoracic and mediastinal disorders) | 55 (55) | 13 (13)
Stomach illness/Nausea/Diarrhea (Injury, poisoning and procedural complications) | 30 (30) | 14 (14)
Pain/Joint Pain/Muscle Aches/ Back Pain (Injury, poisoning and procedural complications) | 23 (23) | 6 (6)
Anxiety/Irritability (Psychiatric disorders) | 7 (7) | 2 (2)
Fatigue/Lethargy (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Increased Heart Rate/Heart Palpitations (Cardiac disorders) | 4 (4) | 2 (2)
Injury: knee/foot (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Hernia (Renal and urinary disorders) | 4 (4) | 0 (0)
Gall bladder surgery (Surgical and medical procedures) | 1 (1) | 2 (2)
Urinary Tract Infection, Bladder problems (Renal and urinary disorders) | 2 (2) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 1 (1)
Elevated Blood Pressure (Cardiac disorders) | 1 (1) | 1 (1)
Ringing in Ears (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1) | 1 (1)
Skin biopsy (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No